CLINICAL TRIAL: NCT05269550
Title: PSMA MRI Guided Prostate SBRT(ARGOS)/Comprehensive, Longitudinal Evaluation of Imaging Biomarkers Post Radiotherapy (CLIMBER)
Brief Title: PSMA MRI Guided Prostate SBRT (ARGOS)/Comprehensive, Longitudinal Evaluation of Imaging Biomarkers Post Radiotherapy (CLIMBER)
Acronym: ARGOS/CLIMBER
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's (Other)
Responsible Party: Principal Investigator, Glenn Bauman, Principle Investigator, London Health Sciences Centre Research Institute OR Lawson Research Institute of St. Joseph's
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ARGOS/CLIMBER
Record Dates: First submitted 2022-01-12; First posted 2022-03-08 (Actual); Last update posted 2025-07-28 (Actual); Status verified 2025-07

CONDITIONS: Prostate Cancer
Keywords: High intermediate risk prostate cancer; High-risk prostate cancer
MeSH Terms: conditions — Prostatic Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Men with high intermediate to very high risk prostate cancer (Experimental): Men with high intermediate to very high risk prostate cancer
  Interventions: Radiation: High-Intermediate Risk Patients-cohort 1; Radiation: High Risk or Very High-Risk Patients-cohort 1; Radiation: High-Intermediate Risk Patients-cohort 2; Radiation: High Risk or Very High-Risk Patients-cohort 2

INTERVENTIONS:
Radiation: High-Intermediate Risk Patients-cohort 1 — Patients will receive 35Gy/5 fractions to the whole prostate (25 Gy to proximal Seminal Vesicles) with a simultaneous boost to PET/MRI defined intra-prostatic foci to a target maximum dose of 50Gy/5 fractions. Six months of androgen deprivation therapy will commence with the end of radiotherapy (concurrent plus adjuvant)
Radiation: High Risk or Very High-Risk Patients-cohort 1 — Patients will receive 35Gy/5 fractions to the whole prostate (25Gy to whole Seminal Vesicles) with a simultaneous boost to PET/MRI defined intra-prostatic foci to a target maximum dose of 50Gy/5 fractions. Pelvic lymph nodes will receive 25Gy/5 fractions synchronous with prostate treatment with a simultaneous boost to imaging involved nodes to a maximum of 35Gy/5 fractions. Eighteen months of androgen deprivation therapy will commence with the end of radiotherapy (concurrent plus adjuvant)
Radiation: High-Intermediate Risk Patients-cohort 2 — Patients will receive 35Gy/5 fractions to the whole prostate (25 Gy to proximal Seminal Vesicles) with a simultaneous boost to PET/MRI defined intra-prostatic foci to a target maximum dose of 50Gy/5 fractions. Androgen deprivation therapy will commence 3 months before radiotherapy (concurrent plus adjuvant) and will continue for a total of 6 months.
Radiation: High Risk or Very High-Risk Patients-cohort 2 — Patients will receive 35Gy/5 fractions to the whole prostate (25 Gy to proximal Seminal Vesicles) with a simultaneous boost to PET/MRI defined intra-prostatic foci to a target maximum dose of 50Gy/5 fractions. Androgen deprivation therapy will commence 3 months before radiotherapy (concurrent plus adjuvant) and will continue for a total of 18 months.

SUMMARY:
This study is a prospective Phase I/II protocol enrolling men with either high intermediate-risk or high-risk or very high-risk prostate cancer. All men will have PSMA Targeted PET (using the PSMA targeting ligand PSMA 1007) and multiparametric magnetic resonance imaging (mpMRI) for delineation of intra-prostatic foci of cancer and any involved regional lymph nodes based on high SUV uptake on PET or mpMRI (T2W, DWI/ADC, DCE) appearance suspicious for cancer. Tumour delineation will be performed by fusing the PSMA PET and mpMRI with planning CT simulation images. Fiducial marker implantation for treatment guidance will be mandatory but use of other organs at risk protection strategies (i.e. GU Loc, Space-OAR) will be allowed but not mandatory. Patients will be treated with image-guided SBRT using the fiducial markers for intra-fraction motion management. Dose escalation to imaging defined targets (intra-prostatic and involved nodes on PSMA PET + MRI) will be accomplished through a simultaneous boost technique. Maintaining dose to organs at risk will take precedence over boost dose targets (targeted maximum dose of 50Gy/5 fractions to imaging defined prostatic lesion; 35Gy/5 fractions to imaging defined involved nodes).

Cohort extension: We hypothesize that integration of neoadjuvant androgen deprivation therapy will provide for pretreatment cancer downstaging and will allow us to achieve higher target doses to the imaging defined DILs than currently achieve. Additionally, we plan to include a novel sodium MRI protocol into the baseline imaging to compare DIL volumes delineated by this modality to those by mpMRI and PSMA PET and to characterize changes in sodium MRI in response to ADT alone and subsequent radiotherapy

ELIGIBILITY:
Inclusion Criteria:

* Age > 18 years of age
* Histologically confirmed carcinoma of the prostate
* High-intermediate risk or high risk as defined by NCCN criteria:
* High intermediate: 2 or 4 intermediate risk factors (T2B-T2C, Gleason GG 2 or 3, PSA 10-20) or GG 3 or intermediate risk with equal or >50% biopsy core involvement
* High-risk: one of T3a, Gleason GG 4 or 5, or PSA >20 ng/ml
* Very-high risk: one of primary Gleason Pattern 5, >4 cores Grade Group 4 or 5, clinical T3b, or more than 1 high-risk feature
* Conventional imaging (bone scan and abdominal pelvic computed tomography) negative for extra-pelvic nodal, skeletal or visceral metastases
* Willing to give informed consent to participate in this clinical trial
* Able and willing to complete EPIC questionnaires

Exclusion Criteria:

* Prior prostate cancer treatment (apart from prior 5-alpha reductase inhibitor treatment); androgen deprivation therapy prior to enrollment or treatment planning not permitted
* Men with clinical T4 disease are excluded
* Contraindication to radical prostate radiotherapy e.g. connective tissue disease or inflammatory bowel disease
* Contraindication to prostate MRI (i.e. non0compatible stent, pacemaker, prosthesis, etc.)
* Contraindication to use of PSMA PET agent PSMA 1007 due to intolerance or allergy
* Anticoagulation medication (if unsafe to discontinue for gold seed insertion)
* Diagnosis of bleeding diathesis
* Poor baseline urinary function defined as a score of 5 ("big problem") on question 5 of the EPIC 26 (Overall, how big a problem has your urinary function been for you during the last 4 weeks?)
* Definitive extra-pelvic nodal or distant metastatic disease on conventional staging investigations

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2022-05-03 (Actual); Primary Completion 2028-12-15 (Estimated); Study Completion 2028-12-15 (Estimated)

PRIMARY OUTCOMES:
6-month Toxicity | 6-months
  6-month gastrointestinal (GI) and genitourinary (GU) toxicity using the Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0).
6-week Toxicity | 6-weeks
  6-week gastrointestinal (GI) and genitourinary (GU) toxicity using the Common Terminology Criteria for Adverse Events version 5.0 (CTCAE v5.0).
Expansion cohort: Median minimum dose to dominant intra-prostatic lesion | 6-months
  Expansion cohort: Median minimum dose to dominant intra-prostatic lesion

SECONDARY OUTCOMES:
Quality of Life measured by the Expanded Prostate Cancer Index Composite (EPIC-26) questionnaires | 5 years
  Quality of life measured by the Expanded Prostate Cancer Index Composite (EPIC-26) questionnaires.
Disease Free Survival | 5 years
  Five-year disease-free survival (DFS) as a composite of biochemical control, patient death or development of clinical metastases or institution of salvage ADT.

OTHER OUTCOMES:
Translational Endpoint 1 | 24 months
  Serial PSMA PET/MRI images will be collected at baseline, 6 months and 2 years to characterize the imaging response of prostate cancer to treatment and potentially identify imaging biomarkers (including pharmacokinetic, radiomic and quantitative PET and mpMRI metrics) that predict for five-year DFS
Translational Endpoint 2 | 24 Months
  Baseline collection of diagnostic tissue biopsy samples and serial collection of blood and urine over multiple time points (baseline, 6 months, 1 year, 2 years post radiotherapy) for correlative biologic biomarker analyses with imaging changes and disease-free survival and toxicity post treatment
Translational Endpoint 3 | 2 years
  A prostate biopsy at baseline and 2 years will allow for correlation of histopathology with PSMA PET/MRI images. Specifically, we will investigate biopsy correlations with pre-treatment PSMA PET/MRI images and whether a negative PSMA PET/MRI is correlated with a negative 2-year post treatment biopsy (shown to correlate with long term disease control
Translational Endpoint 4 | 5 years
  Examine novel clinical prognostic biomarkers (i.e. percentage of Gleason Pattern 4 on biopsy, 4- year PSA response rate) and their correlation with imaging findings and 5-year Disease Free Survival
Translational Endpoint- Expansion cohort | 6 months
  Characterize intra-prostatic foci on pre, post 3-month ADT and 6 months post radiotherapy on PSMA PET/MRI + sodium MRI imaging

CONTACTS AND LOCATIONS:
Locations (2):
- Canada (2):
  - London Health Sciences Centre, London, Ontario
  - Sunnybrook Research Institute, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No